CLINICAL TRIAL: NCT04349293
Title: Ex-vivo Evaluation of the Reactivity of the Immune Infiltrate of Cancers to Treatments With Monoclonal Antibodies Targeting the Immunomodulatory Pathways
Acronym: MAB IN SITRO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2016-A00732-49; 2015/2331 (Other: CSET number)
Record Dates: First submitted 2020-04-14; First posted 2020-04-16 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with cancer (Experimental)
  Interventions: Procedure: Tissue sampling; Procedure: Blood sampling

INTERVENTIONS:
Procedure: Tissue sampling — Collection of a sample of tumor tissue and a sample of adjacent or counter lateral healthy tissue (if possible) from the surgical room
Procedure: Blood sampling — Collection of a 30mL peripheral blood sample in heparin at several times: during surgical and medical treatment (before surgery, before the start of mAbs and after mAbs)

SUMMARY:
Multicentric interventional prospective study with collection of biological samples as part of a routine care research

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years.
2. Male and female sex.
3. Any patient with cancer (see list in the body of the protocol) requiring treatment by surgical resection and / or who will start treatment with mAb or BiTE.
4. Patient information and signed informed consent.
5. Subjects affiliated (or beneficiary) to a social security scheme

Patients treated for immune complications by immunosuppressants may be included (corticosteroids, etc.).

Exclusion Criteria:

1. History of severe systemic autoimmune disease.
2. Pregnant or breastfeeding patient
3. Impossibility or refusal to sign informed consent
4. Patient under guardianship or curatorship, or deprived of liberty by a judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-09-08 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Immunophenotyping of immune infiltrates by flow cytometry | Up yo one year
  Immunophenotyping analysis by flow cytometry (Cyan, Beckman Coulter): identification of several immune sub-populations (T-B-NK lymphocytes, myeloid and tumor cells); identifications of several receptors and ligands (PD1 / PDL1, Tim-3 / HAVCR2,, CTLA-4, 4-1BB / 4-1BBL, Fas / FasL, TRAIL, OX40 / OX40L, ICOS / ICOSL, CD69, CD25 / CD127, NKp46 / NKp30, NKG2D / NKG2DL, galectin-9, MHC class I and II, B7H3 / B7H6); identification of memory subpopulations (CD45RA / CD27 / CCR7) and, if available, intra-cytoplasmic labeling (CXCR3, CCR6, Granzyme B, KI67, TNFα IFNg, IL-17 and IL-21).

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, Val De Marne, France